CLINICAL TRIAL: NCT07242534
Title: Effect of Semaglutide on Embryo Quality in Overweight and Obese Patients Undergoing In Vitro Fertilization. A Randomized Controlled Trial
Brief Title: Effect of Semaglutide on Embryo Quality in Overweight and Obese Patients Undergoing In Vitro Fertilization.
Acronym: SEQ
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion Dexeus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FSD-SEM-2025-14; 2025-522525-34-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Infertility; Obesity
Keywords: Obesity; Overweight; GLP-1 receptor agonist; IVF; ART
MeSH Terms: conditions — Infertility; Obesity; Overweight | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semaglutide (Experimental): Semaglutide 0.25-1.0 mg for 12 weeks prior to ovarian stimulation
  Interventions: Drug: Semaglutide
- No pre-treatment (Active Comparator): No pre-treatment prior to ovarian stimulation Pre-treatment
  Interventions: Other: No pre-treatment

INTERVENTIONS:
Drug: Semaglutide — Participants in this group will receive semaglutide for 12 weeks before ovarian stimulation (0.25 mg/week in weeks 1-4, 0.5 mg/week in weeks 5-8, and 1 mg/week in weeks 9-12). After pre-treatment, controlled ovarian stimulation will be initiated with 225-300 IU/day of rFSH, GnRH antagonist (0.25 mg/day) starting when follicles reach ≥14 mm, and ovulation triggered with triptorelin 0.2 mg when 2-3 follicles reach ≥18 mm. Oocyte retrieval will occur 34-36 hours later, followed by IVF/ICSI. Embryos will be cultured to blastocyst stage and cryopreserved. Embryo transfer will occur after an 8-week washout from semaglutide.
  Arms: Semaglutide
Other: No pre-treatment — Participants in this group will undergo standard ovarian stimulation without semaglutide pre-treatment. Stimulation will begin with 225-300 IU/day of rFSH, GnRH antagonist (0.25 mg/day) starting when follicles reach ≥14 mm, and ovulation triggered with triptorelin 0.2 mg when 2-3 follicles reach ≥18 mm. Oocyte retrieval will be performed 34-36 hours later, followed by IVF/ICSI. Embryos will be cultured to the blastocyst stage and cryopreserved. Embryo transfer will follow standard clinical practice.
  Arms: No pre-treatment

SUMMARY:
This is a randomized, controlled clinical trial with a two-sided superiority hypothesis. The study evaluates whether a 12-week pre-treatment with semaglutide prior to ovarian stimulation improves the number of good-quality blastocysts in overweight and obese women undergoing in vitro fertilization (IVF), compared to no pre-treatment.

DETAILED DESCRIPTION:
Overweight and obese women (BMI 27-40 kg/m²) aged ≤38 years with adequate ovarian reserve (AMH ≥1 ng/mL or AFC ≥6) will be enrolled. Participants will be randomized in a 1:1 ratio to receive either 12 weeks of semaglutide pre-treatment (intervention group) or no pre-treatment (control group) before undergoing standard ovarian stimulation.

Embryos will be cultured to the blastocyst stage and cryopreserved (freeze-all strategy). In the semaglutide group, embryo transfer will occur after an 8-week washout from the last semaglutide dose.

Primary outcome: number of good-quality blastocysts on day 5. Secondary outcomes: embryo morphokinetics, fertilization rate, number of MII oocytes, number of COCs, total blastocyst formation rate, number of cryopreserved embryos, and pre/post semaglutide changes in weight, BMI, waist circumference, AMH, and AFC.

The study has been designed with a superiority hypothesis to detect a difference of 1.5 good-quality blastocysts between groups, with 80% power and a two-sided alpha of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* ≤ 38 years
* AMH >= 1 ng/mL or AFC >= 6
* Body mass index (BMI) between 27 kg/m2 and 40 kg/m2
* Scheduled for IVF with freeze-all strategy

Exclusion Criteria:

* Severe male factor (sperm concentration <5M/mL)
* Type 2 diabetes mellitus
* Prior use of GLP-1 Ras within the past year
* Uncontrolled thyroid disorders
* Contraindications to IVF or semaglutide treatment
* Patients with chronic inflammatory diseases
* Family history of hereditary or chromosomal diseases
* Use of glucocorticoids or immunosuppressants
* PGT-A
* Use of medications affecting metabolism or inflammation

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2026-01-19 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Number of good quality blastocysts (GQB) | Assessed once per participant, from oocyte retrieval (Day 0) to Day 5 of embryo culture, when embryos reach blastocyst stage.
  (ASEBIR criteria

SECONDARY OUTCOMES:
Days of stimulation | From stimulation start (Stimulation Day 1) to trigger day, approx. 8-12 days per participant.
Total dose of Gonadotropins | From first day of ovarian stimulation to trigger day (8-12 days total).
Number COCs | Assessed on day of oocyte retrieval, approx. 34-36 hours after ovulation trigger.
Number MII | Assessed on same day as oocyte retrieval, after denudation and classification
Fertilization rate | Assessed on Day 1 after ICSI, 16-18 hours post-injection
Time of appearance of the 2nd polar body (tPB2) | Recorded via time-lapse system, within first 8 hours post-ICSI (Day 0).
Time of pronuclei appearance (tPNa) | Measured on Day 1 post-ICSI using time-lapse monitoring.
Evaluation of both pronuclei (PN) | Assessed during pronuclear stage on Day 1 post-ICSI.
Time of pronuclei disappearance (tPNf) | Recorded by time-lapse imaging, approx. 20-24 hours post-ICSI.
Time of division from 2 to 8 cells | Tracked continuously via time-lapse, from Day 2 to Day 3 post-ICSI
Time of compaction (tSC) | Tracked by time-lapse imaging on Day 4 post-ICSI
Time of morula (tM) | Recorded by time-lapse on Day 4 post-ICSI.
Time of cavitation (tSB) | Recorded by time-lapse on Day 5 post-ICSI.
Time of full blastulation (tB) | Measured by time-lapse on Day 5 of embryo culture
Total number of day 5 blastocysts | Counted on Day 5 of embryo culture after ICSI
Blastocyst formation rate, | Calculated on Day 5 based on 2PN embryos reaching blastocyst stage.
  the proportion of 2PN zygotes that reach the blastocyst stage
Number of embryos cryopreserved | Recorded at time of freezing on Day 5-7 of embryo culture
Embryo stage (D5, D6, D7) | Assessed at time of embryo cryopreservation on Day 5 to 7
Change in AFC | Compared between baseline (Visit 2) and end of semaglutide treatment (Visit 5, Week 12).
  before and after the treatment with semaglutide
Change in AMH | Compared between baseline (Visit 2) and end of semaglutide treatment (Visit 5, Week 12).
  before and after the treatment with semaglutide
Change in BMI | : Measured at baseline, Weeks 4, 8, and 12 of semaglutide treatment (Visits 2-5).
  before and after the treatment with semaglutide
Change in WC | : Measured at baseline, Weeks 4, 8, and 12 of semaglutide treatment (Visits 2-5).
  before and after the treatment with semaglutide

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos P Polyzos, MD, PhD, Principal Investigator — Dexeus Fertility
Locations (5):
- Spain (5):
  - Dexeus Mujer Sabadell, Sabadell, Barcelona
  - Dexeus Mujer Sant Cugat, Sant Cugat del Vallès, Barcelona
  - Dexeus Mujer Reus, Reus, Tarragona
  - Departamento de Ginecología Obstetricia y Reproducción. Hospital Universitari Dexeus, Barcelona
  - Dexeus Mujer Tarragona, Tarragona

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Amiri M, Ramezani Tehrani F. Potential Adverse Effects of Female and Male Obesity on Fertility: A Narrative Review. Int J Endocrinol Metab. 2020 Sep 28;18(3):e101776. doi: 10.5812/ijem.101776. eCollection 2020 Jul. PMID 33257906
- [Background] Bader S, Bhatti R, Mussa B, Abusanana S. A systematic review of GLP-1 on anthropometrics, metabolic and endocrine parameters in patients with PCOS. Womens Health (Lond). 2024 Jan-Dec;20:17455057241234530. doi: 10.1177/17455057241234530. PMID 38444070
- [Background] Dag ZO, Dilbaz B. Impact of obesity on infertility in women. J Turk Ger Gynecol Assoc. 2015 Jun 1;16(2):111-7. doi: 10.5152/jtgga.2015.15232. eCollection 2015. PMID 26097395
- [Background] Gautam D, Purandare N, Maxwell CV, Rosser ML, O'Brien P, Mocanu E, McKeown C, Malhotra J, McAuliffe FM; FIGO Committee on Impact of Pregnancy on Long-term Health and the FIGO Committee on Reproductive Medicine, Endocrinology and Infertility. The challenges of obesity for fertility: A FIGO literature review. Int J Gynaecol Obstet. 2023 Jan;160 Suppl 1(Suppl 1):50-55. doi: 10.1002/ijgo.14538. PMID 36635080
- [Background] Goldberg AS, Boots CE. Treating obesity and fertility in the era of glucagon-like peptide 1 receptor agonists. Fertil Steril. 2024 Aug;122(2):211-218. doi: 10.1016/j.fertnstert.2024.05.154. Epub 2024 May 27. PMID 38810863
- [Background] He Y, Lu Y, Zhu Q, Wang Y, Lindheim SR, Qi J, Li X, Ding Y, Shi Y, Wei D, Chen ZJ, Sun Y. Influence of metabolic syndrome on female fertility and in vitro fertilization outcomes in PCOS women. Am J Obstet Gynecol. 2019 Aug;221(2):138.e1-138.e12. doi: 10.1016/j.ajog.2019.03.011. Epub 2019 Mar 22. PMID 30910544
- [Background] Jensterle M, Janez A, Fliers E, DeVries JH, Vrtacnik-Bokal E, Siegelaar SE. The role of glucagon-like peptide-1 in reproduction: from physiology to therapeutic perspective. Hum Reprod Update. 2019 Jul 1;25(4):504-517. doi: 10.1093/humupd/dmz019. PMID 31260047
- [Background] Khan D, Ojo OO, Woodward OR, Lewis JE, Sridhar A, Gribble FM, Reimann F, Flatt PR, Moffett RC. Evidence for Involvement of GIP and GLP-1 Receptors and the Gut-Gonadal Axis in Regulating Female Reproductive Function in Mice. Biomolecules. 2022 Nov 23;12(12):1736. doi: 10.3390/biom12121736. PMID 36551163
- [Background] Li MC, Minguez-Alarcon L, Arvizu M, Chiu YH, Ford JB, Williams PL, Attaman J, Hauser R, Chavarro JE; EARTH Study Team. Waist circumference in relation to outcomes of infertility treatment with assisted reproductive technologies. Am J Obstet Gynecol. 2019 Jun;220(6):578.e1-578.e13. doi: 10.1016/j.ajog.2019.02.013. Epub 2019 Feb 11. PMID 30763543
- [Background] Moran L, Tsagareli V, Norman R, Noakes M. Diet and IVF pilot study: short-term weight loss improves pregnancy rates in overweight/obese women undertaking IVF. Aust N Z J Obstet Gynaecol. 2011 Oct;51(5):455-9. doi: 10.1111/j.1479-828X.2011.01343.x. Epub 2011 Jul 19. PMID 21806596
- [Background] Nuako A, Tu L, Reyes KJC, Chhabria SM, Stanford FC. Pharmacologic Treatment of Obesity in Reproductive Aged Women. Curr Obstet Gynecol Rep. 2023 Jun;12(2):138-146. doi: 10.1007/s13669-023-00350-1. Epub 2023 Feb 27. PMID 37427372
- [Background] Pavli P, Triantafyllidou O, Kapantais E, Vlahos NF, Valsamakis G. Infertility Improvement after Medical Weight Loss in Women and Men: A Review of the Literature. Int J Mol Sci. 2024 Feb 5;25(3):1909. doi: 10.3390/ijms25031909. PMID 38339186
- [Background] Sacha CR, Page CM, Goldman RH, Ginsburg ES, Zera CA. Are women with obesity and infertility willing to attempt weight loss prior to fertility treatment? Obes Res Clin Pract. 2018 Jan-Feb;12(1):125-128. doi: 10.1016/j.orcp.2017.11.004. Epub 2017 Dec 6. PMID 29221938
- [Background] Salamun V, Jensterle M, Janez A, Vrtacnik Bokal E. Liraglutide increases IVF pregnancy rates in obese PCOS women with poor response to first-line reproductive treatments: a pilot randomized study. Eur J Endocrinol. 2018 Jul;179(1):1-11. doi: 10.1530/EJE-18-0175. Epub 2018 Apr 27. PMID 29703793
- [Background] Silvestris E, de Pergola G, Rosania R, Loverro G. Obesity as disruptor of the female fertility. Reprod Biol Endocrinol. 2018 Mar 9;16(1):22. doi: 10.1186/s12958-018-0336-z. PMID 29523133
- [Background] Szczesnowicz A, Szeliga A, Niwczyk O, Bala G, Meczekalski B. Do GLP-1 Analogs Have a Place in the Treatment of PCOS? New Insights and Promising Therapies. J Clin Med. 2023 Sep 12;12(18):5915. doi: 10.3390/jcm12185915. PMID 37762856
- [Background] Sola-Leyva A, Pathare ADS, Apostolov A, Aleksejeva E, Kask K, Tammiste T, Ruiz-Duran S, Risal S, Acharya G, Salumets A. The hidden impact of GLP-1 receptor agonists on endometrial receptivity and implantation. Acta Obstet Gynecol Scand. 2025 Feb;104(2):258-266. doi: 10.1111/aogs.15010. Epub 2024 Dec 18. PMID 39696822
- [Background] Sundararaman L, Gouda D, Kumar A, Sundararaman S, Goudra B. Glucagon-like Peptide-1 Receptor Agonists: Exciting Avenues Beyond Weight Loss. J Clin Med. 2025 Mar 14;14(6):1978. doi: 10.3390/jcm14061978. PMID 40142784
- [Background] Wilding JPH, Batterham RL, Calanna S, Davies M, Van Gaal LF, Lingvay I, McGowan BM, Rosenstock J, Tran MTD, Wadden TA, Wharton S, Yokote K, Zeuthen N, Kushner RF; STEP 1 Study Group. Once-Weekly Semaglutide in Adults with Overweight or Obesity. N Engl J Med. 2021 Mar 18;384(11):989-1002. doi: 10.1056/NEJMoa2032183. Epub 2021 Feb 10. PMID 33567185
- See also: Related Info — http://www.dexeus.com